CLINICAL TRIAL: NCT03544502
Title: Is Music the Food of Anesthesia in Children?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Sevtap Hekimoglu Sahin, Clinical Professor, Trakya University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: TUTF-GOKAEK 2013/147; TUTF-GOKAEK (Registry Identifier: Local Ethic)
Record Dates: First submitted 2018-04-11; First posted 2018-06-01 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Music
Keywords: music, anesthesia, surgery
MeSH Terms: interventions — Ear Protective Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music group (Experimental): Music group (group M, n=35) patients applied CD player. One CDs were prepared with 5 children's songs (classic music) for the study. CD player opened during anesthesia induction and continued until postoperative 15 minute
  Interventions: Device: CD player; Device: CEL-480 Sound Level Meter Sonometre
- Silence group (Experimental): silence group (group S, n=35) patients received the independent anesthesiologist applied earplugs into the patients' ears during anesthesia induction and the earplugs were removed immediately before tracheal tube extubation.
  During each measurement, noise level recordings were performed using CEL-480 Sound Level Meter Sonometre.
  Interventions: Device: CEL-480 Sound Level Meter Sonometre; Device: Earplug
- Noise group (Placebo Comparator): noise group (group N, n=35) patients were exposed to the ambient operating room noise.
  Noise level recordings were performed using CEL-480 Sound Level Meter Sonometre.Postoperatively, Emergence delirium (ED) was assessed as a Pediatric Anesthesia Emergence Delirium (PAED) Score ≥ 10.
  Interventions: Device: CEL-480 Sound Level Meter Sonometre; Procedure: Ambient operating room noise

INTERVENTIONS:
Device: CD player — CD player opened during anesthesia induction and continued until postoperative 15 minute
  Other Names: player
  Arms: Music group
Device: CEL-480 Sound Level Meter Sonometre — Noise level recordings were performed using CEL-480 Sound Level Meter Sonometre.
  Other Names: Sonometre
Device: Earplug — the independent anesthesiologist placed earplug into the patients' ears during anesthesia induction and the ear plug were removed immediately before tracheal tube extubation.
  Arms: Silence group
Procedure: Ambient operating room noise — patients were exposed to the ambient operating room noise.
  Arms: Noise group

SUMMARY:
The patients were randomly separated into three groups. Group M (n=35) applied CD player and Group S (n=35) received the independent anesthesiologist placed earplugs into the patients' ears. Group N (n=35) exposed to the ambient operating room noise.

DETAILED DESCRIPTION:
Hundred and five pediatric patients who scheduled for abdominal surgery in ASA I-II risk groups were enrolled in the study. The patients were randomly separated into three groups. Group M (n=35) applied CD player and Group S (n=35) received the independent anesthesiologist placed earplugs into the patients' ears. Group N (n=35) exposed to the ambient operating room noise. The preoperative children's anxiety levels were assessed with the M-YPAS in the operating room. Heart rate (HR) and mid-arterial pressure (MAP) were recorded at 30-minute intervals until the completion of surgery, end of surgery and postoperative. During each measurement, noise level recordings were performed using sonometre. Pediatric Anesthesia Emergence Delirium Score (PEAD) was assessed after extubation, postoperative.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for elective abdominal surgery with an expected operation time of 60 to 120 minutes, were enrolled in the study.

Exclusion Criteria:

* Children were excluded from the study if they had cognitive disorders, with clinically evident hearing impairment, chronic illness, undergoing emergency surgery, and unstable medical conditions requiring intensive care unit admission.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — age from 5 to 9 years of age
Enrollment: 105 (Actual)
Dates: Start 2013-08-28 (Actual); Primary Completion 2015-08-28 (Actual); Study Completion 2016-08-24 (Actual)

PRIMARY OUTCOMES:
Postoperatively, Emergence delirium (ED) was assessed as a Pediatric Anesthesia Emergence Delirium | 15 minutes in postoperative
  Pediatric Anesthesia Emergence Delirium Score was assessed postoperative 15th minutes.

REFERENCES:
- [Derived] Hekimoglu Sahin S, Duran R, Basaran UN, Sut N, Colak A, Duran S. Is music the food of the anesthesia in children? World J Pediatr Surg. 2022 Mar 1;5(2):e000328. doi: 10.1136/wjps-2021-000328. eCollection 2022. PMID 36474510